CLINICAL TRIAL: NCT03287323
Title: The Influence of a Proactive Palliative Care Intervention on Family Satisfaction and Biopsychosocial Problem-related Distress of Patients in a Surgical Intensive Care Unit: A Prospective Single-center Interventional Study
Brief Title: Proactive Palliative Care Intervention in a Surgical ICU: Influence on Family Satisfaction and Patient Distress
Acronym: PALL-ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Rita Laufenberg-Feldmann, M.D., Anaesthesiologist, Head of Clinical Trial Unit, Johannes Gutenberg University Mainz
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 837.108.17 (10942)
Record Dates: First submitted 2017-09-08; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Palliative Care
Keywords: palliative care; surgical intensive care; family satisfaction; ICU decision-making; end-of-life care

STUDY DESIGN:
Intervention Model Description: Prospective before-and after interventional study including 100 patients who receive usual intensive care followed by an interventional part with 100 patients who receive additional palliative care consultations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): One hundred patients of a control group will receive standard intensive care treatment (Usual Care Group).
- Proactive Palliative Care (Other): One hundred patients will additionally be offered a palliative care Intervention (Proactive Palliative Care Group).
  Interventions: Other: Proactive Palliative Care

INTERVENTIONS:
Other: Proactive Palliative Care — In the intervention part of the study, enrolled patients will be offered a set of different palliative care interventions, including symptom management, advance care planning, palliative physiotherapy, social and spiritual support, communication with patients and caregivers, in addition to standard intensive care.
  Arms: Proactive Palliative Care

SUMMARY:
Patients will be identified according to pre-defined trigger criteria for a palliative intervention. One hundred patients of a control group will receive standard intensive care treatment (Usual Care Group). Patients' biopsychosocial problem-related distress will be evaluated and family satisfaction with intensive care will be measured with standardized questionnaires. In the subsequent intervention part of the study one hundred patients will additionally be offered a palliative care treatment (Proactive Care Group) and patients' biopsychosocial problem-related distress as well as family satisfaction will also be evaluated.

DETAILED DESCRIPTION:
The project consists of different consecutive parts:

1. Trigger criteria: Trigger criteria for patients with unmet palliative care needs in an intensive care unit have been specified prior to start of the clinical study by survey of staff of the surgical intensive care unit (intensivists and nursing staff): Trigger criteria include a) advanced cancer, b) multi-organ failure, c) severe cognitive impairment or dementia
2. Clinical study: Proactive palliative care intervention vs. standard care for intensive care patients. Initially patients fulfilling the defined trigger criteria will be enrolled in the standard care group (Group 1). In the intervention part of the study, enrolled patients will be offered a set of different palliative care interventions in addition to standard intensive care (Group 2). In both groups, family satisfaction will be evaluated with the FS-ICU-24 (Family Satisfaction Intensive Care) questionnaire after discharge of the patients from the ICU. 8 weeks (60 days +/- 7 days) after inclusion in the study, patients' biopsychosocial distress will be assessed with standardized patient questionnaires (NCCN Distress thermometer, PHQ-2 Patient Health Questionnaire). One year after inclusion in the study, patients' functional status will be evaluated in a telephone interview using the Barthel Index. Planned duration of clinical part of the study: 3 years, thereof

   1. Patient-related:

      Duration of palliative care intervention: approx. 60 mins for each patient contact. The number of interventions depends on the duration of ICU stay per patient. Follow-up per patient until 1 year after enrolment.
   2. Study-related:

   The clinical study starts with the enrollment of the first ICU patient. Data will be collected between the admission of the patient in the ICU until discharge from ICU and hospital discharge, respectively. Follow-up visits will be performed 8 weeks and 1 year after enrolment. Patients will be recruited over an estimated period of approx. 3 years, assuming that 1-2 patients per week can be included. Follow-up data will be collected up to 1 year after last patient in.
3. Termination of study including data analysis and evaluation, and publication of the study results: approx. 1 year

ELIGIBILITY:
Inclusion Criteria:

* need for intensive care for more than 3 days and at least one of the following trigger criteria:

  1. known advanced cancer
  2. severe cognitive impairment or dementia
  3. multi-organ failure

Exclusion Criteria:

* Patients who already receive palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
family satisfaction in a surgical intensive care unit using a standardized questionnaire (FS-ICU). | after discharge from ICU, up to 1 year after enrolment
  To evaluate the effects of a proactive palliative care intervention for selected patients with unmet palliative needs on family satisfaction in a surgical intensive care unit using a standardized questionnaire (FS-ICU).

SECONDARY OUTCOMES:
Patients' biopsychosocial problem-related distress after intensive care treatment measured with the NCCN distress thermometer | 60 days +/- 7 days after enrolment
  To evaluate the effects of a proactive palliative care intervention for selected patients with unmet palliative needs in a surgical intensive care unit on patients' self-reported distress, measured with the NCCN distress thermometer
Intensive care length of stay | up to 1 year after enrolment
  To evaluate the effects of a proactive palliative care intervention for selected patients with unmet palliative needs in a surgical intensive care unit on ICU length of stay, measured as days in ICU.
Duration of hospitalization | up to 1 year after enrolment
  To evaluate the effects of a proactive palliative care intervention for selected patients with unmet palliative needs in a surgical intensive care unit on hospital length of stay, measured as days in hospital.
1-year Patient survival | up to 1 year after enrolment
  To evaluate the effects of a proactive palliative care intervention for selected patients with unmet palliative needs in a surgical intensive care unit on overall survival of patients.
Organ replacement therapy | up to 1 year after enrolment
  To evaluate organ dysfunction and duration of replacement therapy, measured as days of mechanical ventilation and/or days of ECMO and/or days of hemofiltration, if applicable
Functional assessment after 1 year | up to 1 year after enrolment
  To evaluate functionality with regard to activities of daily living (Barthel Index)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, University Medical Center of Johannes Gutenberg-University Mainz, Germany, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hua M, Wunsch H. Integrating palliative care in the ICU. Curr Opin Crit Care. 2014 Dec;20(6):673-80. doi: 10.1097/MCC.0000000000000149. PMID 25233330
- [Result] Heyland DK, Tranmer JE; Kingston General Hospital ICU Research Working Group. Measuring family satisfaction with care in the intensive care unit: the development of a questionnaire and preliminary results. J Crit Care. 2001 Dec;16(4):142-9. doi: 10.1053/jcrc.2001.30163. PMID 11815899
- [Result] Wall RJ, Engelberg RA, Downey L, Heyland DK, Curtis JR. Refinement, scoring, and validation of the Family Satisfaction in the Intensive Care Unit (FS-ICU) survey. Crit Care Med. 2007 Jan;35(1):271-9. doi: 10.1097/01.CCM.0000251122.15053.50. PMID 17133189
- [Result] Selecky PA, Eliasson CA, Hall RI, Schneider RF, Varkey B, McCaffree DR; American College of Chest Physicians. Palliative and end-of-life care for patients with cardiopulmonary diseases: American College of Chest Physicians position statement. Chest. 2005 Nov;128(5):3599-610. doi: 10.1378/chest.128.5.3599. PMID 16304319
- [Result] Mosenthal AC, Weissman DE, Curtis JR, Hays RM, Lustbader DR, Mulkerin C, Puntillo KA, Ray DE, Bassett R, Boss RD, Brasel KJ, Campbell M, Nelson JE. Integrating palliative care in the surgical and trauma intensive care unit: a report from the Improving Palliative Care in the Intensive Care Unit (IPAL-ICU) Project Advisory Board and the Center to Advance Palliative Care. Crit Care Med. 2012 Apr;40(4):1199-206. doi: 10.1097/CCM.0b013e31823bc8e7. PMID 22080644
- [Result] Braus N, Campbell TC, Kwekkeboom KL, Ferguson S, Harvey C, Krupp AE, Lohmeier T, Repplinger MD, Westergaard RP, Jacobs EA, Roberts KF, Ehlenbach WJ. Prospective study of a proactive palliative care rounding intervention in a medical ICU. Intensive Care Med. 2016 Jan;42(1):54-62. doi: 10.1007/s00134-015-4098-1. Epub 2015 Nov 10. PMID 26556622